CLINICAL TRIAL: NCT05149066
Title: #KindGirlsInACTion: A School-based Intervention to Promote Compassive Competences and Psychological Flexibility in Female Adolescents
Brief Title: #KindGirlsInACTion: A Programme for the Promotion of Mental Health of Female Adolescents
Acronym: KindGirlsACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Joana Marta-Simões (Unknown)
Responsible Party: Principal Investigator, Ana Laura Mendes, Integrated non-PhD member of CINEICC, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #KindGirlsInACTion
Record Dates: First submitted 2021-11-15; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Quality of Life; Eating Disorders; Eating Behavior; Psychological; Emotion Regulation; Body Image; Relations, Interpersonal
Keywords: Intervention Programme; School-based; Adolescence; Girls; Psychological well-being; Compassion; Psychological flexibility; Positive body image
MeSH Terms: conditions — Feeding and Eating Disorders; Feeding Behavior; Emotional Regulation; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group was administered a 9-sessions weekly programme in the school context.
  It completed three assessment moments: pre-intervention, post-intervention and a 3-months after the intervention follow-up.
  Interventions: Behavioral: #KindGirlsInACTion
- Control group (No Intervention): The control group did not receive any intervention. It completed three assessment moments: pre-intervention, post-intervention and a 3-months after the intervention follow-up.

INTERVENTIONS:
Behavioral: #KindGirlsInACTion — 9-session weekly cognitive-behavioural intervention to promote psychological well-being and prevent body image and eating-related disordered behaviours.
  Arms: Experimental group

SUMMARY:
The #KindGirlsInACTion project started in 2017 and developed and implemented a psychotherapeutic intervention program in Portuguese female adolescents. This program aimed to improve the overall quality of life and well-being of the participants, and specifically to promote a qualitative improvement in body image and interpersonal relationships, through the promotion of self-compassion, compassion and psychological flexibility. #KindGirlsInACTion is a school-based program, with 9 sessions over 9 weeks. It is essentially practical and interactive, with exercises created specifically for the program, as well as the regular practice of mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* being a female adolescent;
* being aged between 12 and 18;
* being a part of a classroome with immediate availability to attend the sessions.

Exclusion Criteria:

* Having a clinical condition that could compromise the completion of self-report questionnaires;
* Having a significant score on screening measures administered pre-intervention.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Psychological Well-being | 5 months
  Kidscreen-27
Psychological Well-being | 3 months
  Kidscreen-27
Psychological Wel--being | Baseline
  Kidscreen-27

SECONDARY OUTCOMES:
Eating Disorders | Baseline
  Eating Disorders Examination Questionnaire, EDE-Q
Eating Disorders | 3 months
  Eating Disorders Examination Questionnaire, EDE-Q
Eating Disorders | 5 months
  Eating Disorders Examination Questionnaire, EDE-Q
Positive body image | Baseline
  Body Appreciation Scale, BAS-2
Positive body image | 3 months
  Body Appreciation Scale, BAS-2
Positive body image | 5 months
  Body Appreciation Scale, BAS-2
Social safeness | Baseline
  Social Safeness and Pleasure Scale, SSPS
Social safeness | 3 months
  Social Safeness and Pleasure Scale, SSPS
Social safeness | 5 months
  Social Safeness and Pleasure Scale, SSPS
Body image shame | Baseline
  Body Image Shame Scale, BISS
Body image shame | 3 months
  Body Image Shame Scale, BISS
Body image shame | 5 months
  Body Image Shame Scale, BISS

CONTACTS AND LOCATIONS:
Locations (1):
- CINEICC, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No